CLINICAL TRIAL: NCT07345182
Title: Lower Dislocation But Higher Fracture Risk: Posterior vs. Lateral Approaches in Hemiarthroplasty for Femoral Neck Fractures
Brief Title: Clinical and Functional Outcomes of Lateral vs Posterior Hemiarthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Yusuf Bayram, Orthopaedic Surgeon, Umraniye Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B.10.1.TKH.4.34.H.GP.0.01/91
Record Dates: First submitted 2025-12-23; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Femoral Neck Fractures; Hip Fractures; Hemiarthroplasty
Keywords: Lateral Hemiarthroplasty; Posterior Hemiarthroplasty; Surgical Approach; Functional Outcome; Harris Hip Score; Parker and Palmer Mobility Score
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned in a 1:1 ratio to one of two parallel groups to undergo hemiarthroplasty using either the lateral or the posterior surgical approach. Each participant received only the assigned intervention.
Masking Description: This study was conducted as an open-label trial. Due to the nature of the surgical interventions, blinding of surgeons and participants was not feasible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral Approach Group (Experimental): Patients underwent hemiarthroplasty using the direct lateral surgical approach.
  Interventions: Procedure: Lateral approach hemiarthroplasty
- Posterior Approach Group (Experimental): Patients underwent hemiarthroplasty using the posterior surgical approach.
  Interventions: Procedure: Posterior approach hemiarthroplasty

INTERVENTIONS:
Procedure: Posterior approach hemiarthroplasty — Hemiarthroplasty performed using the posterior surgical approach.
  Arms: Posterior Approach Group
Procedure: Lateral approach hemiarthroplasty — Hemiarthroplasty performed using the lateral surgical approach.
  Arms: Lateral Approach Group

SUMMARY:
This prospective, single-center, randomized clinical trial compared the clinical and functional outcomes of hemiarthroplasty performed via lateral versus posterior surgical approaches in elderly patients with displaced intracapsular femoral neck fractures. The primary objective was to compare prosthetic dislocation and intraoperative femoral fracture rates between the two approaches. Secondary outcomes included functional scores, radiological parameters, complications, and mortality.

DETAILED DESCRIPTION:
This study is a prospective, single-center, randomized clinical trial designed to compare the clinical, functional, and radiological outcomes of hemiarthroplasty performed via lateral and posterior surgical approaches in elderly patients with displaced intracapsular femoral neck fractures.

Between March 2016 and June 2019, eligible patients were randomized in a 1:1 ratio to undergo hemiarthroplasty using either the lateral or posterior approach. Randomization was performed using a computer-generated sequence. All procedures were performed or supervised by experienced orthopedic surgeons following standardized surgical and postoperative protocols.

Clinical parameters, perioperative data, and radiological indices including cortical index, Singh index, and Dorr classification were recorded. Functional outcomes were assessed using the Parker and Palmer Mobility Score (PPMS) and the Harris Hip Score (HHS). Patients were followed for a minimum of 12 months.

The primary outcome measure was the prosthetic dislocation rate within 12 months postoperatively. Secondary outcomes included intraoperative periprosthetic femoral fracture rate, functional scores, complications, and mortality. The study was conducted in accordance with the principles of the Declaration of Helsinki, with approval obtained from the local ethics committee, and written informed consent was obtained from all participants or their legal representatives.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* Displaced intracapsular femoral neck fracture
* Treated with hemiarthroplasty
* Ability to provide informed consent by the patient or a legal representative

Exclusion Criteria:

* Pathological femoral neck fractures
* Previous surgery on the affected hip
* Polytrauma patients
* Periprosthetic fractures

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Prosthetic dislocation rate | Within 12 months postoperatively
  Incidence of postoperative prosthetic hip dislocation following hemiarthroplasty.

SECONDARY OUTCOMES:
Intraoperative periprosthetic femoral fracture rate | During surgery
  Incidence of intraoperative femoral fractures occurring during hemiarthroplasty.
Harris Hip Score (HHS) | Preoperative baseline and final follow-up at minimum 12 months postoperatively
  The Harris Hip Score is a clinician-based outcome measure ranging from 0 to 100 points, where higher scores indicate better hip function.
Parker and Palmer Mobility Score (PPMS) change | Preoperative baseline and final follow-up at minimum 12 months postoperatively
  The Parker and Palmer Mobility Score is a validated mobility assessment scale ranging from 0 to 9 points, where higher scores indicate better mobility.
One-year mortality | Within 12 months postoperatively
  All-cause mortality within one year after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Ümraniye Training and Research Hospital, Istanbul, Umraniye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.